CLINICAL TRIAL: NCT06565624
Title: Evaluation of Reflex Tear Production
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Management decision post planned futility analysis
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DEF512-E004
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Dry Eye Disease
Keywords: Reflex Tear Production
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nasal Stimulation (Experimental): The Investigator will insert cotton swabs into both nostrils of the subject and gently probe the nasal middle cavities. Stimulation will stop once visible and obvious reflex tearing has begun.
  Interventions: Procedure: Cotton Swab Nasal Stimulation

INTERVENTIONS:
Procedure: Cotton Swab Nasal Stimulation — Nostril probing for the purpose of producing reflex tearing

SUMMARY:
The purpose of this study is to evaluate reflex tear production following cotton swab nasal stimulation in subjects with dry eye disease (DED).

DETAILED DESCRIPTION:
The primary analysis will assess the change from baseline (pre- versus immediately post-cotton swab nasal stimulation) in tear meniscus height (TMH) using optical coherence tomography (OCT). This study will consist of one visit on a single day.

ELIGIBILITY:
Key Inclusion Criteria:

* Within the last 12 months, have a previous history of dry eye disease, either clinician diagnosed or patient reported.
* Within the last 6 months, have used, or desired to use artificial tears for dry eye symptoms.
* Corrected Visual Acuity (Snellen) 20/200 or better in both eyes.
* Good general and ocular health, as determined by the investigator using medical history, ophthalmic examination and history.
* Able, as assessed by the investigator, and willing to follow study instructions.
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Current evidence of any clinically significant ophthalmic disease other than dry eye (for example, glaucoma or macular degeneration).
* Use of artificial tears within 2 hours of the Study Visit.
* History of ocular surgery within 1 year of the Study Visit.
* Use of contact lenses in either eye within 7 days of the Study Visit.
* Use of lid hygiene (all forms of lid care) or heat masks within 7 days of the Study Visit.
* Use of any topical ocular anti-inflammatory medications, any topical ocular corticosteroid, or any non-steroidal-anti-inflammatory agents within 30 days of the Study Visit.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-10-17 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in TMH immediately following stimulation | Day 1 pre-stimulation (Baseline); Day 1 immediately post-stimulation
  TMH (the distance between the line of reflection along the top of the tear prism to the edges of the eyelids) will be measured in millimeters using OCT, a non-invasive imaging test that uses light waves to take cross-section pictures of the eye. TMH will be assessed prior to nasal stimulation and upon completion of nasal stimulation. Only one eye will be assessed by OCT.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Pharma, Study Director — Alcon Research, LLC
Locations (1):
- Eye Research Foundation, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No